CLINICAL TRIAL: NCT03444584
Title: An Exploratory Phase 2a Randomized, Placebo-controlled, Double-blind Study to Evaluate the Efficacy and Safety of MEDI0382 Versus Placebo in Overweight/Obese Subjects With Type 2 Diabetes Mellitus Treated With Dapagliflozin and Metformin
Brief Title: Study of MEDI0382 in Combination With Dapagliflozin and Metformin in Overweight/Obese Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5670C00007; 2017-002817-78 (EudraCT Number)
Record Dates: First submitted 2017-10-18; First posted 2018-02-23 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: 0382; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cotadutide; Metformin

STUDY DESIGN:
Intervention Model Description: Efficacy and Safety of MEDI0382 versus Placebo in Overweight/Obese Participants with Type 2 Diabetes Mellitus Treated with Dapagliflozin and Metformin
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, Placebo-controlled, Double-blind Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MEDI0382 (Experimental): Participants will receive subcutaneous dose of MEDI0382 daily (titrated up from 100 μg for 7 days to 200 μg for 7 days and to 300 μg for 14 days) for 28 days. Participants were on metformin and dapagliflozin background dual therapy during the treatment period.
  Interventions: Drug: MEDI0382; Drug: Dapaglifozin; Drug: Metformin
- Placebo (Placebo Comparator): Participants will receive subcutaneous dose of placebo matched to MEDI0382 daily for 28 days. Participants were on metformin and dapagliflozin background dual therapy during the treatment period
  Interventions: Drug: Placebo; Drug: Dapaglifozin; Drug: Metformin

INTERVENTIONS:
Drug: MEDI0382 — Subcutaneous dose of MEDI0382 (titrated up from 100 μg for 7 days to 200 μg for 7 days and to 300 μg for 14 days).
  Arms: MEDI0382
Drug: Placebo — Subcutaneous dose of placebo matched to MEDI0382.
  Arms: Placebo
Drug: Dapaglifozin — Oral dose of dapaglifozin 10 mg tablet.
Drug: Metformin — Oral dose of metformin tablet (maximum tolerated dose [MTD] > 1 g).

SUMMARY:
A Phase 2 study Comparing the effects on glucose control of MEDI0382 in combination with Dapagliflozin and Metformin compared to placebo in combination with Dapagliflozin and Metformin in overweight/obese participants with Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
This is an exploratory randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of MEDI0382 versus placebo in overweight/obese participants with T2DM treated with metformin and dapagliflozin dual therapy. The study will enroll participants with T2DM treated either with metformin monotherapy or with metformin and dapagliflozin dual therapy. After the screening period, participants treated with metformin monotherapy only will enter a 4-week run-in period where participants will be administered oral dapagliflozin 10 mg a day, which will be provided by the sponsor. Enrolled participants that are already treated with metformin and dapagliflozin dual therapy will continue this dual therapy throughout the study and can be randomized after the screening period without entering the run-in period. All participants (ie, on monotherapy and dual therapy) entering the double-blind treatment period will receive dapagliflozin 10 mg a day, which will be provided by the sponsor.

Participants in this study will participate for up to 20 weeks including a screening period of up to 60 days, a 4-week run-in period (for participants on metformin monotherapy only), a 4-week treatment period, and a 4-week follow-up post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged >= 18 years at screening.
2. Provision of signed and dated informed consent form (ICF) prior to any study specific procedures.
3. Body mass index between 25 kg/m^2 and 40 kg/m^2 (inclusive) at screening.
4. Hemoglobin A1c range between 7.0% and 10.0% (inclusive) at the time of screening.
5. Diagnosed with T2DM and treated with of metformin monotherapy (MTD > 1 g) at least 8 weeks prior to screening or treated with stable, oral doses of dapagliflozin 10 mg and metformin (MTD > 1 g) for at least 3 months prior screening.
6. Participants prescribed oral dual therapy with sulphonylurea, glitinide, or dipeptidyl peptidase-4 inhibitor (in addition to metformin) may be eligible to enter the study following a washout period of these medications totaling at least 28 days before initial screening evaluations have been completed.
7. Participants treated with stable doses of metformin (MTD > 1 g) with canagliflozin (maximum dose of 300 mg/day), or metformin (MTD > 1 g) with empaglifozin (maximum dose of 25mg/day) for at least 3 months prior to screening may be eligible to enter the study after switching to dapagliflozin.
8. Female participants of childbearing potential must have a negative pregnancy test at screening and randomization and must not be lactating.
9. Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception from screening and must agree to continue using such precautions through to the end of the study. It is strongly recommended for the male partner of a female participant to also use male condom plus spermicide throughout this period. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.

Exclusion Criteria:

1. History of, or any existing condition that in the opinion of the investigator would interfere with evaluation of the investigational product, put the participant at risk, influence the participant's ability to participate, or affect the interpretation of the results of the study and/or any participant unable or unwilling to follow study procedures.
2. Any participant who has received another investigational product not included in the protocol as part of a clinical trial or a glucagon-like peptide-1 (GLP-1) analogue or sodium-glucose cotransporter-2 (SGLT2)-containing preparation (excluding dapagliflozin, canagliflozin, empagliflozin) within the last 30 days or 5 half-lives of the drug (whichever is longest) at the time of screening.
3. Any participant who has received any of the following medications prior to the start of the screening period (Visit 1) or prior to the study start period (Visit 4):

   * Concurrent use of any medicinal products, or herbal or over-the-counter (OTC) preparations licensed for control of body weight or appetite at the time of screening (Visit 1)
   * Concurrent or previous use of drugs approved for weight loss (eg, orlistat, bupropion-naltrexone, phentermine-topiramate, phentermine, lorcaserin) within the last 30 days or 5 half-lives of the drug (whichever is longest) at the time of screening (Visit 1)
   * Concurrent use of aspirin (acetylsalicylic acid) at a dose greater than 150 mg once daily and within the last 72 hours prior to the start of the study (Visit 4)
   * Concurrent use of paracetamol (acetaminophen) or paracetamol-containing preparations at a total daily dose of greater than 3000 mg and within the last 72 hours prior to the start of the study (Visit 4)
   * Concurrent use of ascorbic acid (vitamin C) supplements at a total daily dose greater than 1000 mg and within the last 72 hours prior to the start of the study (Visit 4)
   * Concurrent use of opiates, domperidone, metoclopramide, or other drugs known to alter gastric emptying and within the last 72 hours prior to the start of the study (Visit 4)
4. Concurrent participation in another study of any kind and repeat randomization in this study is prohibited.
5. Severe allergy/hypersensitivity to any of the proposed study treatments or excipients.
6. Diagnosis of type 1 diabetes mellitus, maturity-onset diabetes of the young, or latent autoimmune diabetes of adulthood or presence of anti-glutamic acid decarboxylase, anti-islet cell, or anti-insulin antibodies.
7. Symptoms of acutely decompensate blood glucose control (eg, thirst, polyuria, weight loss) at screening or randomization, a history of diabetes ketoacidosis (DKA), or hyperosmolar nonketotic coma or treatment with daily subcutaneous insulin within 90 days prior to screening.
8. Fasting hyperglycemia (> 250 mg/dL/ > 13.9 mmol/L) prior to randomization.
9. C-peptide level < lower limit of normal (LLN).
10. History of acute or chronic pancreatitis or pancreatectomy.
11. Hypertriglyceridemia (> 400 mg/dL) at screening.
12. Significant inflammatory bowel disease, gastroparesis, or other severe disease or surgery affecting the upper gastrointestinal (GI) tract (including weight-reducing surgery and procedures) which may affect gastric emptying or could affect the interpretation of safety and tolerability data.
13. Significant hepatic disease (except for nonalcoholic steatohepatitis or nonalcoholic fatty liver disease without portal hypertension or cirrhosis) and/or participants with any of the following results at screening:

    * Aspartate transaminase (AST) >= 3 × upper limit of normal (ULN)
    * Alanine transaminase (ALT) >= 3 × ULN
    * Total bilirubin (TBL) >= 2 × ULN
14. Impaired renal function defined as estimated glomerular filtration rate (eGFR) <= 60 mL/minute/1.73m^2 at screening (eGFR according to Modification of Diet in Renal Disease [MDRD] using the isotope dilution mass spectrometry-traceable MDRD Study Equation (SI units).
15. Use of loop diuretics within 1 month prior to screening.
16. Poorly controlled hypertension as defined below:

    * Systolic blood pressure (BP) > 160 mm Hg
    * Diastolic BP or >= 100 mm Hg After 10 minutes of supine rest and confirmed by repeated measurement at screening (Visit 1 for all participants).
17. Unstable angina pectoris, myocardial infarction, transient ischemic attack, or stroke within 3 months prior to screening, or participants who have undergone percutaneous coronary intervention or a coronary artery bypass graft within the past 6 months or who are due to undergo these procedures at the time of screening.
18. Severe congestive heart failure (New York Heart Association Class III and IV)
19. Basal calcitonin level > 50 ng/L at screening or history/family history of medullary thyroid carcinoma or multiple endocrine neoplasia.
20. Hemoglobinopathy, hemolytic anemia, or chronic anemia (hemoglobin concentration < 11.5 g/dL [115 g/L] for males and < 10.5 g/dL [105 g/L] for females) at screening or any other condition known to interfere with interpretation of HbA1c measurement.
21. History of neoplastic disease within 5 years prior to screening, except for adequately treated basal cell skin cancer, squamous cell skin cancer, or in situ cervical cancer.
22. Any positive results for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus antibody.
23. Recent viral infection or illness requiring the use of antibiotics in the month prior to screening (Visit 1) for participants on dual therapy or prior to run-in period (Visit 2) for participants on monotherapy.
24. History of recurrent (at least 2) urinary tract and/or genital tract infections (including mycotic infections such as thrush) within 6 months prior to screening.
25. Substance dependence likely to impact participant safety or compliance with study procedures.
26. Involvement of any AstraZeneca, MedImmune, contract research organization, or study site employees and their close relatives.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bain, MD, Principal Investigator — Joint Clinical Research Facility
Locations (8):
- Germany (3):
  - Research Site, Magdeburg
  - Research Site, Mannheim
  - Research Site, München
- Hungary (3):
  - Research Site, Balatonfüred
  - Research Site, Miskolc
  - Research Site, Szeged
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Rotherham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: D5670C00007-Clinical-Protocol draft Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00007&attachmentIdentifier=7da0c75e-9474-4771-b53c-2ba877a1f0db&fileName=D5670C00007-Clinical-Protocol_draft_MM_(002)_Redacted.pdf&versionIdentifier=
- See also: D5670C00007 Statistical Analysis Plan Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00007&attachmentIdentifier=78bc8436-d4a9-47f9-b04d-004c6cc68f9e&fileName=D5670C00007_Statistical_Analysis_Plan_redaction_draft_MM_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Germany and Hungary between 08May2018 and 06Dec2018.
Groups:
- Placebo: Participants received subcutaneous dose of placebo matched to MEDI0382 daily for 28 days. Participants were on metformin and dapagliflozin background dual therapy during the treatment period.
- MEDI0382: Participants received subcutaneous dose of MEDI0382 daily (titrated up from 100 μg for 7 days to 200 μg for 7 days and to 300 μg for 14 days) for 28 days. Participants were on metformin and dapagliflozin background dual therapy during the treatment period.
Period: Overall Study
Arm/Group | Placebo | MEDI0382
Started | 24 | 25
Completed | 24 | 23
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any dose of study drugs and analyzed according to the treatment they actually received.
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | Placebo | MEDI0382 | TOTAL
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (10.0) | 61.0 (8.2) | 59.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 12 | 15 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 25 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 25 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 28 in Plasma Glucose Area Under the Concentration Time-curve From Time 0 to 4 Hours (AUC0-4hrs) as Measured by Mixed-meal Tolerance Test (MMTT)
Description: The MMTT test involved the consumption of a standardised liquid meal (nutritional supplement of fat, carbohydrate, and protein) within 5 minutes. On Day -1 and on Day 28, following a minimum 10 hour fast, serial of blood samples were obtained prior and through 240 minutes after consumption of standardized meal for the measurement of glucose metabolism (with no additional food intake during this time).
Time Frame: Zero minutes before and 15, 30, 45, 60, 90, 120, 180, and 240 minutes after consumption of the standardised meal on Day -1 (Baseline) and Day 28
Population: Intent-to-treat (ITT) population included all participants who received any dose of study drugs analyzed according to their randomized treatment group. Here, number of participants analyzed "N" signifies participants who were analyzed for the specified outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: hr·mg/dL
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 22 | 24
hr·mg/dL | -11.28 [-51.05 to 28.50] | -154.37 [-192.45 to -116.29]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -143.09, 95% CI 2-sided [-198.20 to -87.98]

2. Primary Outcome: Percent Change From Baseline to Day 28 in Plasma Glucose AUC0-4hrs as Measured by MMTT
Description: The MMTT test involved the consumption of a standardised liquid meal (nutritional supplement of fat, carbohydrate, and protein)within 5 minutes. On Day -1 and on Day 28, following a minimum 10-hour fast, serial of blood samples were obtained prior and through 240 minutes after consumption of standardized meal for the measurement of glucose metabolism (with no additional food intake during this time).
Time Frame: as for outcome 1
Population: An ITT population included all participants who received any dose of study drugs and analyzed according to their randomized treatment group. Here, number of participants analyzed "N" signifies participants who were analyzed for the specified outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change in Glucose AUC0-4hrs
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 22 | 24
Percent change in Glucose AUC0-4hrs | -0.13 [-5.96 to 5.69] | -22.30 [-27.88 to -16.73]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -22.17, 95% CI 2-sided [-30.24 to -14.10]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience(immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 28 days after the last dose of MEDI0382 (approximately 8 weeks)
Population: As-treated population included all participants who received any dose of study drug and analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Participants
  TEAEs | 14 | 13
  TESAEs | 0 | 0

4. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Reported as TEAEs
Description: Number of participants with abnormal 12-lead ECG reported as TEAEs are reported.
Time Frame: Day 1 through 28 days after the last dose of MEDI0382 (approximately 8 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Number of participants with abnormal vital signs reported as TEAEs are reported.
Time Frame: Day 1 through 28 days after the last dose of MEDI0382 (approximately 8 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Participants
  Tachycardia | 2 | 1
  Tachycardia paroxysmal | 1 | 0
  Palpitations | 0 | 1

6. Secondary Outcome: Number of Participants With Abnormal Physical Examinations Reported as TEAEs
Description: Number of participants with abnormal physical examinations reported as TEAEs are reported.
Time Frame: Day 1 through 28 days after the last dose of MEDI0382 (approximately 8 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported.
Time Frame: Day 1 through 28 days after the last dose of MEDI0382 (approximately 8 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Participants
  Hypoglycemia | 1 | 0

8. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC [0-∞]) of MEDI0382
Description: Area under the plasma concentration time curve from time zero to infinity (AUC [0-∞]) of MEDI0382 is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days 7, 14, and 28
Population: MEDI0382 pharmacokinetic (PK) population included all participants who received at least 1 dose of MEDI0382 and had at least 1 MEDI0382 PK sample above the lower limit of quantitation. Here, number analyzed "n" signifies participants who were analyzed for the specified day.
Measure: Geometric Mean (Full Range); unit: ng.hr/mL
Arm/Group | MEDI0382
Number analyzed (Participants) | 25
ng.hr/mL
  Day 7 (MEDI0382 100 µg): number analyzed (Participants) | 9
  Day 7 (MEDI0382 100 µg) | 106.4 [57.7 to 251.8]
  Day 14 ( MEDI0382 200 µg): number analyzed (Participants) | 9
  Day 14 ( MEDI0382 200 µg) | 196.7 [99.4 to 472.0]
  Day 28 (MEDI0382 300 µg): number analyzed (Participants) | 9
  Day 28 (MEDI0382 300 µg) | 314.6 [211.0 to 537.3]

9. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC [0-∞]) of Dapagliflozin
Description: Area under the plasma concentration time curve from time zero to infinity (AUC [0-∞]) of Dapagliflozin is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days -1, 7, 14, and 28
Population: Dapagliflozin PK population included all participants who received at least 1 dose of dapagliflozin and had at least 1 dapagliflozin PK sample above the lower limit of quantitation. Here, number analyzed "n" signifies participants who were analyzed for the specified day.
Measure: Geometric Mean (Full Range); unit: ng.hr/mL
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
ng.hr/mL
  Day -1: number analyzed (Participants) | 20 | 24
  Day -1 | 432.6 [271.5 to 918.6] | 473.8 [288.8 to 1073.2]
  Day 7: number analyzed (Participants) | 15 | 12
  Day 7 | 410.2 [209.9 to 1024.2] | 438.0 [222.2 to 833.6]
  Day 14: number analyzed (Participants) | 16 | 8
  Day 14 | 421.0 [219.0 to 1327.8] | 448.6 [247.0 to 615.9]
  Day 28: number analyzed (Participants) | 15 | 16
  Day 28 | 405.7 [261.1 to 799.5] | 523.4 [319.5 to 946.0]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve During the Dosing Period (AUCtau) of MEDI0382
Description: Area under the plasma concentration-time curve during the dosing period (AUCtau) of MEDI0382 is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days 7, 14, and 28
Population: MEDI0382 PK population included all participants who received at least 1 dose of MEDI0382 and had at least 1 MEDI0382 PK sample above the lower limit of quantitation. Here, number analyzed "n" signifies participants who were analyzed for the specified day.
Measure: Geometric Mean (Full Range); unit: ng.hr/mL
Arm/Group | MEDI0382
Number analyzed (Participants) | 25
ng.hr/mL
  Day 7 (MEDI0382 100 µg): number analyzed (Participants) | 23
  Day 7 (MEDI0382 100 µg) | 89.6 [43.1 to 199.4]
  Day 14 ( MEDI0382 200 µg): number analyzed (Participants) | 23
  Day 14 ( MEDI0382 200 µg) | 165.0 [86.9 to 365.5]
  Day 28 (MEDI0382 300 µg): number analyzed (Participants) | 22
  Day 28 (MEDI0382 300 µg) | 265.9 [101.7 to 795.1]

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve During the Dosing Period (AUCtau) of Dapagliflozin
Description: Area under the plasma Concentration-time curve during the dosing period (AUCtau) of Dapagliflozin is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days -1, 7, 14, and 28
Population: as for outcome 9
Measure: Geometric Mean (Full Range); unit: ng.hr/mL
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
ng.hr/mL
  Day -1: number analyzed (Participants) | 24 | 24
  Day -1 | 400.9 [182.4 to 1011.5] | 430.3 [252.5 to 815.2]
  Day 7 | 377.5 [76.4 to 910.7] | 406.8 [211.5 to 1142.6]
  Day 14: number analyzed (Participants) | 23 | 23
  Day 14 | 417.1 [209.0 to 1107.7] | 396.8 [215.4 to 669.7]
  Day 28: number analyzed (Participants) | 23 | 24
  Day 28 | 423.1 [180.6 to 977.3] | 463.8 [284.3 to 1245.7]

12. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI0382
Description: Maximum observed serum concentration (Cmax) of MEDI0382 is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days 7, 14, and 28
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | MEDI0382
Number analyzed (Participants) | 25
ng/mL
  Day 7 (MEDI0382 100 µg) | 5.2 [2.7 to 11.9]
  Day 14 ( MEDI0382 200 µg): number analyzed (Participants) | 24
  Day 14 ( MEDI0382 200 µg) | 10.1 [4.4 to 21.7]
  Day 28 (MEDI0382 300 µg): number analyzed (Participants) | 22
  Day 28 (MEDI0382 300 µg) | 17.2 [6.1 to 45.4]

13. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Dapagliflozin
Description: Maximum observed serum concentration (Cmax) of Dapagliflozin is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days -1, 7, 14, and 28
Population: as for outcome 9
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
ng/mL
  Day -1 | 110.1 [46.3 to 208.3] | 116.7 [38.2 to 206.8]
  Day 7 | 92.0 [5.2 to 256.7] | 84.4 [24.1 to 211.7]
  Day 14: number analyzed (Participants) | 23 | 24
  Day 14 | 95.6 [33.5 to 280.7] | 61.1 [15.8 to 149.9]
  Day 28: number analyzed (Participants) | 23 | 24
  Day 28 | 112.2 [47.0 to 235.4] | 94.2 [25.2 to 182.2]

14. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of MEDI0382
Description: Time to reach maximum observed serum concentration (Tmax) of MEDI0382 is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days 7, 14, and 28
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | MEDI0382
Number analyzed (Participants) | 25
Hours
  Day 7 (MEDI0382 100 µg) | 5.5 [2 to 8]
  Day 14 ( MEDI0382 200 µg): number analyzed (Participants) | 24
  Day 14 ( MEDI0382 200 µg) | 5.1 [2 to 8]
  Day 28 (MEDI0382 300 µg): number analyzed (Participants) | 22
  Day 28 (MEDI0382 300 µg) | 4 [1.9 to 8.1]

15. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of Dapagliflozin
Description: Time to reach maximum observed serum concentration (Tmax) of Dapagliflozin is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days -1, 7, 14, and 28
Population: as for outcome 9
Measure: Median (Full Range); unit: Hours
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Hours
  Day -1 | 1 [0.5 to 2] | 1 [0.4 to 23.9]
  Day 7 | 1 [0.5 to 11.4] | 1 [0.5 to 4]
  Day 14: number analyzed (Participants) | 23 | 24
  Day 14 | 1.1 [0.5 to 6] | 1 [0 to 8.1]
  Day 28: number analyzed (Participants) | 23 | 24
  Day 28 | 1 [0.2 to 1.8] | 1 [0.5 to 8.1]

16. Secondary Outcome: Terminal Elimination Half-life (t½) of MEDI0382
Description: Terminal half-life is the time required for the plasma concentration to fall by 50% during the terminal phase. The t½ of MEDI0382 is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days 7, 14, and 28
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: Hours
Arm/Group | MEDI0382
Number analyzed (Participants) | 25
Hours
  Day 7 (MEDI0382 100 µg): number analyzed (Participants) | 9
  Day 7 (MEDI0382 100 µg) | 8.8 [6.1 to 11.9]
  Day 14 ( MEDI0382 200 µg): number analyzed (Participants) | 9
  Day 14 ( MEDI0382 200 µg) | 9 [5.6 to 11.8]
  Day 28 (MEDI0382 300 µg): number analyzed (Participants) | 9
  Day 28 (MEDI0382 300 µg) | 9.1 [5.1 to 11.6]

17. Secondary Outcome: Terminal Elimination Half-life (t½) of Dapagliflozin
Description: Terminal half-life is the time required for the plasma concentration to fall by 50% during the terminal phase. The t½ of Dapagliflozin is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days -1, 7, 14, and 28
Population: as for outcome 9
Measure: Geometric Mean (Full Range); unit: Hours
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Hours
  Day -1: number analyzed (Participants) | 20 | 24
  Day -1 | 8.2 [5.3 to 11.2] | 7.8 [5.4 to 11.3]
  Day 7: number analyzed (Participants) | 15 | 12
  Day 7 | 7.9 [4.1 to 10.4] | 8.3 [5.8 to 11.1]
  Day 14: number analyzed (Participants) | 16 | 8
  Day 14 | 7.0 [5.1 to 11.4] | 8.5 [7 to 10]
  Day 28: number analyzed (Participants) | 15 | 16
  Day 28 | 7.6 [5.8 to 11.0] | 9.1 [6.1 to 11.8]

18. Secondary Outcome: Apparent Clearance (CL/F) of MEDI0382
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. The CL/F of MEDI0382 is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days 7, 14, and 28
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: L/hr
Arm/Group | MEDI0382
Number analyzed (Participants) | 25
L/hr
  Day 7 (MEDI0382 100 µg): number analyzed (Participants) | 9
  Day 7 (MEDI0382 100 µg) | 1.1 [0.5 to 1.9]
  Day 14 ( MEDI0382 200 µg): number analyzed (Participants) | 9
  Day 14 ( MEDI0382 200 µg) | 1.3 [0.5 to 2.2]
  Day 28 (MEDI0382 300 µg): number analyzed (Participants) | 9
  Day 28 (MEDI0382 300 µg) | 1.2 [0.8 to 1.8]

19. Secondary Outcome: Apparent Clearance (CL/F) of Dapagliflozin
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. The CL/F of Dapagliflozin is reported.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hrs post-dose on Days -1, 7, 14, and 28
Population: as for outcome 9
Measure: Geometric Mean (Full Range); unit: L/Hr
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
L/Hr
  Day -1: number analyzed (Participants) | 20 | 24
  Day -1 | 25.5 [13.3 to 38.9] | 23.3 [12.3 to 39.6]
  Day 7: number analyzed (Participants) | 15 | 12
  Day 7 | 26.7 [11.0 to 52.8] | 25.7 [14.2 to 47.3]
  Day 14: number analyzed (Participants) | 16 | 8
  Day 14 | 25.9 [9.0 to 47.7] | 25.5 [18.8 to 46.4]
  Day 28: number analyzed (Participants) | 15 | 16
  Day 28 | 26.8 [13.8 to 40.2] | 22.2 [13.4 to 35.2]

20. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) Titer to MEDI0382
Description: Number of participants with positive Anti-drug antibodies (ADA) titer to MEDI0382 are reported.
Time Frame: Day 1 (pre-dose), on Day 29 , and 28 days post last dose (end of study visit; approximately 8 weeks)
Population: Immunogenicity population included all participants who received any dose of study drug (MEDI0382 or placebo) and analyzed according to the treatment they actually received and had at least one serum sample for immunogenicity testing. Here, number analyzed "n" signifies participants who were analyzed for the specified day.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Participants
  Day 1 | 0 | 3
  Day 29: number analyzed (Participants) | 24 | 24
  Day 29 | 0 | 1
  End of Study: number analyzed (Participants) | 24 | 24
  End of Study | 1 | 2

21. Secondary Outcome: Change From Baseline in Plasma Glucose AUC24-hrs to the End of Each Dosing Level as Measured by Continuous Glucose Monitoring (CGM)
Description: Continuous glucose monitoring is a minimally invasive device applied to the skin in the upper arm that provides a measure of interstitial glucose levels every 15 minutes. Continuous glucose monitoring measures glucose excursions during different meals and at different times of the day. End of dosing: Day 7 for MEDI0382 100 μg; Day 14 for MEDI0382 200 μg; and Day 28 for MEDI0382 300 μg.
Time Frame: Day -1 (Baseline) through Day 7 for MEDI0382 100 μg, Day 14 for MEDI0382 200 μg, and Day 28 for MEDI0382 300 μg
Population: An ITT population included all participants who received any dose of study drug (MEDI0382 or placebo) and analyzed according to their randomized treatment group. Here, number analyzed "n" signifies participants who were analyzed for the specified day.
Measure: Mean (Standard Deviation); unit: hr.mg/dL
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
hr.mg/dL
  Day 7 (MEDI0382 100 μg): number analyzed (Participants) | 10 | 12
  Day 7 (MEDI0382 100 μg) | 49.14 (667.30) | -832.66 (506.22)
  Day 14 (MEDI0382 200 μg): number analyzed (Participants) | 9 | 13
  Day 14 (MEDI0382 200 μg) | 57.30 (379.95) | -666.05 (647.63)
  Day 28 (MEDI0382 300 μg): number analyzed (Participants) | 12 | 18
  Day 28 (MEDI0382 300 μg) | 229.47 (589.19) | -726.85 (710.71)

22. Secondary Outcome: Change From Baseline in Mean 24-hrs Plasma Glucose to the End of Each Dosing Level as Measured by CGM
Description: as for outcome 21
Time Frame: Day -1 (Baseline) through Day 7 for MEDI0382 100 μg, Day 14 for MEDI0382 200 μg, and Day 28 for MEDI0382 300 μg
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
mg/dL
  Day 7 (MEDI0382 100 μg): number analyzed (Participants) | 10 | 12
  Day 7 (MEDI0382 100 μg) | 2.59 (28.96) | -34.74 (20.34)
  Day 14 (MEDI0382 200 μg): number analyzed (Participants) | 9 | 13
  Day 14 (MEDI0382 200 μg) | 2.83 (17.01) | -28.34 (27.12)
  Day 28 (MEDI0382 300 μg): number analyzed (Participants) | 12 | 18
  Day 28 (MEDI0382 300 μg) | 9.70 (24.73) | -30.55 (29.82)

23. Secondary Outcome: Change From Baseline in Standard Deviation of 24-hrs Plasma Glucose Readings to the End of Each Dosing Level as Measured by CGM
Description: as for outcome 21
Time Frame: Day -1 (Baseline) through Day 7 for MEDI0382 100 μg, Day 14 for MEDI0382 200 μg, and Day 28 for MEDI0382 300 μg
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
mg/dL
  Day 7 (MEDI0382 100 μg): number analyzed (Participants) | 10 | 12
  Day 7 (MEDI0382 100 μg) | -3.01 (13.84) | -7.21 (11.05)
  Day 14 (MEDI0382 200 μg): number analyzed (Participants) | 9 | 13
  Day 14 (MEDI0382 200 μg) | 1.38 (9.47) | -7.52 (9.73)
  Day 28 (MEDI0382 300 μg): number analyzed (Participants) | 12 | 18
  Day 28 (MEDI0382 300 μg) | -4.39 (10.67) | -9.76 (10.18)

24. Secondary Outcome: Change From Baseline in Coefficient of Variation of 24-hrs Plasma Glucose Readings to the End of Each Dosing Level as Measured by CGM
Description: as for outcome 21
Time Frame: Day -1 (Baseline) through Day 7 for MEDI0382 100 μg, Day 14 for MEDI0382 200 μg, and Day 28 for MEDI0382 300 μg
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percent of coefficient of variation
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Percent of coefficient of variation
  Day 7 (MEDI0382 100 μg): number analyzed (Participants) | 10 | 12
  Day 7 (MEDI0382 100 μg) | -2.37 (9.06) | -0.45 (6.68)
  Day 14 (MEDI0382 200 μg): number analyzed (Participants) | 9 | 13
  Day 14 (MEDI0382 200 μg) | 0.96 (8.74) | -2.06 (6.59)
  Day 28 (MEDI0382 300 μg): number analyzed (Participants) | 12 | 18
  Day 28 (MEDI0382 300 μg) | -4.26 (7.16) | -3.21 (7.25)

25. Secondary Outcome: Change From Baseline in Mean Amplitude of Glucose Excursions (MAGE) of 24-hrs Plasma Glucose Readings to the End of Each Dosing Level as Measured by CGM
Description: as for outcome 21
Time Frame: Day -1 (Baseline) through Day 7 for MEDI0382 100 μg, Day 14 for MEDI0382 200 μg, and Day 28 for MEDI0382 300 μg
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
mg/dL
  Day 7 (MEDI0382 100 μg): number analyzed (Participants) | 10 | 12
  Day 7 (MEDI0382 100 μg) | -13.46 (32.07) | -25.74 (35.06)
  Day 14 (MEDI0382 200 μg): number analyzed (Participants) | 9 | 13
  Day 14 (MEDI0382 200 μg) | 18.05 (47.60) | -26.59 (25.60)
  Day 28 (MEDI0382 300 μg): number analyzed (Participants) | 12 | 18
  Day 28 (MEDI0382 300 μg) | -8.09 (27.68) | -27.92 (23.17)

26. Secondary Outcome: Change From Baseline in the Percentage of 24-hrs Glucose Readings That Falls Within the Euglycemic Range to the End of Each Dosing as Measured by CGM
Description: Continuous glucose monitoring is a minimally invasive device applied to the skin in the upper arm that provides a measure of interstitial glucose levels every 15 minutes. Continuous glucose monitoring measures glucose excursions during different meals and at different times of the day. End of dosing: Day 7 for MEDI0382 100 μg; Day 14 for MEDI0382 200 μg; and Day 28 for MEDI0382 300 μg. Euglycemic range is defined as glucose levels of >= 70 mg/dL (>= 3.9 mmol/L) and <= 180 mg/dL (<= 10.0 mmol/L).
Time Frame: Day -1 (Baseline) through Day 7 for MEDI0382 100 μg, Day 14 for MEDI0382 200 μg, and Day 28 for MEDI0382 300 μg
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percent of Euglycemic Range
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Percent of Euglycemic Range
  Day 7 (MEDI0382 100 μg): number analyzed (Participants) | 10 | 12
  Day 7 (MEDI0382 100 μg) | -5.61 (19.65) | 7.12 (20.60)
  Day 14 (MEDI0382 200 μg): number analyzed (Participants) | 9 | 13
  Day 14 (MEDI0382 200 μg) | -2.79 (10.16) | 5.31 (17.71)
  Day 28 (MEDI0382 300 μg): number analyzed (Participants) | 12 | 18
  Day 28 (MEDI0382 300 μg) | -4.17 (15.80) | 6.54 (24.37)

27. Secondary Outcome: Change From Baseline in the Percentage of 24-hrs Glucose Readings That Falls Within the Hyperglycemic Range to the End of Each Dosing as Measured by CGM
Description: Continuous glucose monitoring is a minimally invasive device applied to the skin in the upper arm that provides a measure of interstitial glucose levels every 15 minutes. Continuous glucose monitoring measures glucose excursions during different meals and at different times of the day. End of dosing: Day 7 for MEDI0382 100 μg; Day 14 for MEDI0382 200 μg; and Day 28 for MEDI0382 300 μg. Hyperglycemic (high glucose) range is defined as glucose levels of > 180 mg/dL (> 10.0 mmol/L).
Time Frame: Day -1 (Baseline) through Day 7 for MEDI0382 100 μg, Day 14 for MEDI0382 200 μg, and Day 28 for MEDI0382 300 μg
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percent of hyperglycemic range
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Percent of hyperglycemic range
  Day 7 (MEDI0382 100 μg): number analyzed (Participants) | 10 | 12
  Day 7 (MEDI0382 100 μg) | 3.62 (17.80) | -13.99 (14.95)
  Day 14 (MEDI0382 200 μg): number analyzed (Participants) | 9 | 13
  Day 14 (MEDI0382 200 μg) | 0.36 (10.50) | -9.81 (13.68)
  Day 28 (MEDI0382 300 μg): number analyzed (Participants) | 12 | 18
  Day 28 (MEDI0382 300 μg) | 6.08 (16.96) | -9.72 (20.97)

28. Secondary Outcome: Change From Baseline in the Percentage of 24-hrs Glucose Readings That Falls Within the Hypoglycemic Range to the End of Each Dosing as Measured by CGM
Description: Continuous glucose monitoring is a minimally invasive device applied to the skin in the upper arm that provides a measure of interstitial glucose levels every 15 minutes. Continuous glucose monitoring measures glucose excursions during different meals and at different times of the day. End of dosing: Day 7 for MEDI0382 100 μg; Day 14 for MEDI0382 200 μg; and Day 28 for MEDI0382 300 μg. Hypoglycemic range is defined as glucose levels of < 70 mg/dL (< 3.9 mmol/L).
Time Frame: Day -1 (Baseline) through Day 7 for MEDI0382 100 μg, Day 14 for MEDI0382 200 μg, and Day 28 for MEDI0382 300 μg
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percent of hypoglycemic range
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Percent of hypoglycemic range
  Day 7 (MEDI0382 100 μg): number analyzed (Participants) | 10 | 12
  Day 7 (MEDI0382 100 μg) | 1.17 (5.64) | 6.08 (10.36)
  Day 14 (MEDI0382 200 μg): number analyzed (Participants) | 9 | 13
  Day 14 (MEDI0382 200 μg) | 2.00 (3.79) | 3.44 (12.72)
  Day 28 (MEDI0382 300 μg): number analyzed (Participants) | 12 | 18
  Day 28 (MEDI0382 300 μg) | -2.08 (4.14) | 2.84 (12.20)

29. Secondary Outcome: Change From Baseline in the Percentage of 24-hrs Glucose Readings That Falls Within Clinically Significant Hypoglycemic Range to the End of Each Dosing as Measured by CGM
Description: Continuous glucose monitoring is a minimally invasive device applied to the skin in the upper arm that provides a measure of interstitial glucose levels every 15 minutes. Continuous glucose monitoring measures glucose excursions during different meals and at different times of the day. End of dosing: Day 7 for MEDI0382 100 μg; Day 14 for MEDI0382 200 μg; and Day 28 for MEDI0382 300 μg. Clinically significant hypoglycemic range is defined as glucose levels of < 54 mg/dL (3.0 mmol/L).
Time Frame: Day -1 (Baseline) through Day 7 for MEDI0382 100 μg, Day 14 for MEDI0382 200 μg, and Day 28 for MEDI0382 300 μg
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percent of hypoglycemic range
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 24 | 25
Percent of hypoglycemic range
  Day 7 (MEDI0382 100 μg): number analyzed (Participants) | 10 | 12
  Day 7 (MEDI0382 100 μg) | 0.76 (3.64) | 1.61 (5.03)
  Day 14 (MEDI0382 200 μg): number analyzed (Participants) | 9 | 13
  Day 14 (MEDI0382 200 μg) | 0.27 (1.19) | -0.06 (2.18)
  Day 28 (MEDI0382 300 μg): number analyzed (Participants) | 12 | 18
  Day 28 (MEDI0382 300 μg) | -0.26 (0.90) | 0.93 (4.91)

ADVERSE EVENTS:
Time Frame: Day 1 through 28 days after the last dose of MEDI0382 (approximately 8 weeks)
Arm/Group | Placebo | MEDI0382
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 14/24 | 13/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | MEDI0382 (N=25)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4) | 5 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (6)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (3)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Food craving (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT03444584/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT03444584/SAP_001.pdf